CLINICAL TRIAL: NCT06279728
Title: Medical Access Program for Datopotamab Deruxtecan (Dato-DXd, DS-1062a)
Brief Title: Medical Access Program for Datopotamab Deruxtecan in EGFRm NSCLC Patients
Status: Approved for marketing | Type: Expanded Access
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: DS1062-0003-EAP-MA
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: EGFRm Advanced Non-Small Cell Lung Cancer; EGFRm Metastatic Non-Small Cell Lung Cancer
Keywords: Dato-DXd; Datopotamab; Datapotamab deruxtecan; Deruxtecan; DS-1062a; Named patient program; Emergency use; Compassionate use; Expanded access program; Medical access program; EGFRm Advanced Non-Small Cell Lung Cancer; EGFRm Metastatic Non-Small Cell Lung Cancer; EGFR mutation; EGFR; Mutation

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Datopotamab deruxtecan — 6 mg/kg intravenous infusion Q3W (on Day 1 of each 21-day cycle)
  Other Names: Dato-DXd; DS-1062a

SUMMARY:
The purpose of this Medical Access Program (also referred to as an Expanded Access Program in the USA) is to provide access to Dato-DXd for eligible patients with previously treated advanced or metastatic EGFR mutated non-small cell lung cancer (NSCLC) who, in their treating physician's opinion, have an unmet clinical need, are unlikely to obtain optimal benefit from currently approved and commercially available drugs, and who cannot enter a suitable clinical trial.

DETAILED DESCRIPTION:
This is a Medical Access Program that will be available to adult patients with previously treated advanced or metastatic EGFR mutated NSCLC who have no suitable treatment options and are not able to enter a clinical trial.

Patients enrolled in the Medical Access Program can continue treatment until any of the following occurs:

* Disease progression
* Unacceptable toxicity
* The benefit-risk no longer favors the individual
* Dato-DXd becomes commercially available and reimbursement is approved
* The patient chooses to discontinue treatment
* Withdrawal of consent
* Pregnancy
* Physician discretion
* Death

Patients enrolled in the Medical Access Program have an option to participate in collection of safety-focused clinical practice data. This will contribute towards better understanding of the clinical experience of treatment with Dato-DXd. Participation in this optional data collection will have no bearing on receipt of treatment.

ELIGIBILITY:
Patients are only eligible after signing the informed consent form and must meet all of the following criteria to be eligible for the Medical Access Program.

Inclusion Criteria:

* Patientsis aged ≥18 years (follow local regulatory requirements if the legal age of consent for participation is >18 years old).
* The patient has histologically or cytologically documented advanced or metastatic NSCLC that is not amenable to curative surgery or radiation.
* The patient must have documented AGAs in EGFR (for example, Ex19del, L858R, G719X, S768I or L861Q, either alone or in combination with other EGFR mutations, which may include T790M). Overexpression of EGFR in the absence of activating mutation is not sufficient for enrollment.
* The patient must have progressed on at least 1 EGFR tyrosine kinase inhibitor and platinum-based chemotherapy, either combined or in either sequence.
* The patient has adequate bone marrow reserve and organ function, based on local laboratory data, in the opinion of the treating physician.
* If the patient is a female and of childbearing potential, a negative urine or serum pregnancy test is required at time of treatment initiation request.
* If the patient (male and female) is of reproductive/childbearing potential, they must agree to use a highly effective form of contraception or avoid intercourse during the program and upon completion of this program and for at least 7 months for females and 4 months for males after the last dose of Dato-DXd.
* Starting at the first dose of Dato-DXd, the patient agrees that if they are:

  * A male patient, they must not freeze or donate sperm at any time during this program and for at least 4 months after the last dose of Dato-DXd. Preservation of sperm should be considered prior to the first dose of Dato-DXd.
  * A female patient, they must not donate, or retrieve for their own use, ova at any time during this program and for at least 7 months after the last dose of Dato-DXd. Preservation of ova should be considered prior to the first dose of Dato-DXd.
* The patient must have a life expectancy of >3 months as determined by the treating physician.
* The patient is willing and able to provide written informed consent indicating that they understand the purpose of the Medical Access Program and are willing and able to participate.

Patients who meet any of the following criteria will not be eligible for the Medical Access Program.

Exclusion Criteria:

* The patient has a history of non-infectious ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or have suspected ILD/pneumonitis that cannot be ruled out by imaging at the time of entering the program.
* The patient has clinically severe respiratory compromise (based on treating physician assessment) resulting from intercurrent pulmonary illnesses including, but not limited to:

  * Any underlying pulmonary disorder (e.g., pulmonary emboli within 3 months prior to program enrollment, severe asthma, severe chronic obstructive pulmonary disease, moderate to severe restrictive lung disease, or moderate to severe pleural effusion).
  * Any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement (e.g., rheumatoid arthritis, Sjogren's syndrome, sarcoidosis), OR
  * Prior complete pneumonectomy.
* Patient has clinically significant unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, Grade >1 at start of treatment within the program. Patients with chronic Grade 2 toxicities may be eligible at the discretion of the treating physician after consultation with the Sponsor Medical Approvers or designees within this program.
* Patient has active or uncontrolled hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
* Patient has active hepatitis C. (Active hepatitis C is defined by a positive Hep C Ab result, quantitative HCV ribonucleic acid (RNA) results greater than the lower limits of detection of the assay, and an ALT or AST greater than or equal to 2 times the upper limit of normal.)
* Patient has uncontrolled hepatitis B. (Patients with hepatitis B [positive HBs antigen test] must meet the following criteria to be eligible: have an HBV-DNA viral load <2000 IU/mL off treatment or have an HBV-DNA viral load <2000 IU/mL on oral antiviral therapy for at least 4 weeks and during the participation in the study.)
* The patient has known human immunodeficiency virus (HIV) infection that is not well controlled. All of the following criteria are required to define an HIV infection that is well controlled:

  * Undetectable viral RNA.
  * Cluster of differentiation 4 (CD4)+ count ≥350.
  * No history of acquired immunodeficiency syndrome-defining opportunistic infection within the past 12 months, and stable for at least 4 weeks on the same anti-HIV medications (meaning there are no expected further changes in that time to the number or type of antiretroviral drugs in the regimen).
  * If an HIV infection meets the above criteria, monitoring of viral RNA load and CD4+ count is recommended. Patients must be tested for HIV during the screening period if acceptable by local regulations or an institutional review board (IRB)/ethics committee (EC).
* The patient has a history of severe hypersensitivity reactions to either the drug or inactive ingredients (including but not limited to polysorbate 80) of Dato-DXd.
* The patient has a history of severe hypersensitivity reactions to other monoclonal antibodies.
* Female patient who is pregnant, breast-feeding, or intending to become pregnant.
* The patient has prior or ongoing clinically relevant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the treating physician's opinion, could affect the safety of the patient if prescribed Dato-DXd.
* The patient has clinically significant corneal disease.
* The patient is currently participating in or is in active follow-up (as defined by the protocol) for any Daiichi Sankyo or Astra Zeneca clinical study.
* The patient is eligible for any available oncology clinical trial.
* The patient has received a prior DNA topoisomerase 1 inhibitor (including as a payload of an ADC).
* The patient has received prior radiotherapy to the brain within 2 weeks of start of Dato-DXd treatment or received radiotherapy to the chest within 4 weeks of start of Dato-DXd treatment, or the patient has ongoing radiation-related toxicities requiring corticosteroids.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Affairs, Study Director — Daiichi Sankyo
Locations (14):
- United States (14):
  - Highlands Oncology Group, Springdale, Arkansas
  - Queen's Medical Center, Honolulu, Hawaii
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Touro Infirmary - LCMC Health, New Orleans, Louisiana
  - University of Maryland Medical Center Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Karmanos Cancer Institute (Barbara Ann Karmanos Cancer Hospital), Detroit, Michigan
  - Henry Ford Health, Detroit, Michigan
  - Central Care Cancer Center, Bolivar, Missouri
  - Overlook Medical Center Medical Diagnostic Associates Atlantic Medical Group, Summit, New Jersey
  - New York Cancer & Blood Specialists, New York, New York
  - Baptist Cancer Center, Memphis, Tennessee
  - University of Texas Southwestern Medical, Dallas, Texas
  - Houston Methodist Hospital Cancer Center, Houston, Texas
  - Northwest Medical Specialties, PLLC, Tacoma, Washington